CLINICAL TRIAL: NCT06109831
Title: An Efficacy, Safety Study to Evaluate Multiple Subcutaneous SHR-1918 in Combination With Lipid-Lowering Drugs for the Stable Treatment of Hyperlipidemic Patients With Poor Lipid Control-A Multicenter, Randomized, Double-Blind, Placebo-Parallel-Controlled, Phase II Clinical Study
Brief Title: Evaluate the Efficacy and Safety of SHR-1918 in Patients With Hyperlipidemic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Suncadia Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1918-201
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemic

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase II Clinical Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1918 (Experimental)
  Interventions: Drug: SHR-1918
- SHR-1918 placebo (Placebo Comparator)
  Interventions: Drug: SHR-1918 placebo

INTERVENTIONS:
Drug: SHR-1918 — SHR-1918
  Arms: SHR-1918
Drug: SHR-1918 placebo — SHR-1918 placebo
  Arms: SHR-1918 placebo

SUMMARY:
This is a Multicenter, Randomized, Double-Blind, Placebo-Parallel-Controlled, Phase II Clinical Stud to assess the reduction of low-density lipoprotein cholesterol (LDL-C) by SHR-1918 in patients with Hyperlipidemic.

ELIGIBILITY:
Inclusion Criteria:

1. Regularly taking any moderate-intensity or higher dose* of statin stabilization therapy for ≥4 weeks at screening:

   1. ASCVD risk is ultra-high risk Fasting LDL-C ≥ 1.4 mmol/L;
   2. ASCVD risk very high risk Fasting LDL-C ≥1.8 mmol/L;
   3. ASCVD risk is intermediate or high risk Fasting LDL-C ≥ 2.6 mmol/L.
2. Any other condition that is not met at screening Regularly taking any moderate intensity and higher dose* statin stabilization therapy for ≥4 weeks;

   a) Fasting LDL-C ≥ 2.6 mmol/L.
3. Fasting triglycerides ≤ 5.6 mmol/L.

Exclusion Criteria:

1. Previously diagnosed type 1 diabetes or poorly controlled type 2 diabetes at screening (HbA1c > 8.5%).
2. eGFR <30ml/min/1.73m2 at the screening visit.
3. CK >5times ULN at the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-04 (Actual)

PRIMARY OUTCOMES:
Percent change in calculated LDL-C from baseline to week 16 | from baseline to week 16

SECONDARY OUTCOMES:
Change in calculated LDL-C from baseline to week 16 | from baseline to week 16

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xie X, Shi X, Zhang Y, Su S, Jiang C, Miao L, Wang J, Peng D, Lv L, Chai X, Luo S, Zheng Y, Huang S, Zhu D, Liao S, Ren M, Gao X, Yang H, Zhou H, He Y, Han Y, Xu J, Zhang L, Du L, Yao Z, Sheng J, Peng X, Chen X, Li J, Mi J, Lu Q, Wang H, Shen Z, Zhao Z, Gao F, Lv C, Zhu M, Zhu Y, Wang J. Angiopoietin-Like 3 Antibody Therapy in Patients With Suboptimally Controlled Hyperlipidemia: A Phase 2 Study. J Am Coll Cardiol. 2025 May 20;85(19):1821-1835. doi: 10.1016/j.jacc.2025.03.008. Epub 2025 Mar 31. PMID 40167414